CLINICAL TRIAL: NCT06008717
Title: A Prospective, Randomized Feasibility Clinical Trial Evaluating Bilateral Stimulation of the Dorsolateral Region of the Subthalamic Nucleus Receiving Hyperdirect (M1/SMA) Input in Subjects With Early-Stage Parkinson's Disease
Brief Title: Double-Blind Clinical Trial of Subthalamic Nucleus Deep Brain Stimulation in Early-Stage Parkinson's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mallory Hacker (Other)
Responsible Party: Sponsor-Investigator, Mallory Hacker, Assistant Professor of Neurology, Vanderbilt University Medical Center
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: G220314
Record Dates: First submitted 2022-12-23; First posted 2023-08-24 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: motor scores will be blindly rated by an independent movement disorders neurologist who will be unaware of treatment assignment, ON vs OFF treatment status, or visit sequence
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- active subthalamic nucleus deep brain stimulation plus optimal drug therapy (Experimental): active subthalamic nucleus deep brain stimulation; plus optimal drug therapy
  Interventions: Device: active subthalamic nucleus deep brain stimulation plus optimal drug therapy
- inactive subthalamic nucleus deep brain stimulation plus optimal drug therapy (Active Comparator): inactive subthalamic nucleus deep brain stimulation plus optimal drug therapy
  Interventions: Device: inactive subthalamic nucleus deep brain stimulation plus optimal drug therapy

INTERVENTIONS:
Device: active subthalamic nucleus deep brain stimulation plus optimal drug therapy — active subthalamic nucleus deep brain stimulation (DBS) plus optimal drug therapy
  Arms: active subthalamic nucleus deep brain stimulation plus optimal drug therapy
Device: inactive subthalamic nucleus deep brain stimulation plus optimal drug therapy — optimal drug therapy alone with DBS device turned off
  Arms: inactive subthalamic nucleus deep brain stimulation plus optimal drug therapy

SUMMARY:
The goal of this trial is to evaluate the preliminary safety and efficacy of programming to maximize stimulation of the dorsolateral region of the subthalamic nucleus (STN) receiving primary motor (M1) and supplementary motor area (SMA), but not pre-SMA, input deep brain stimulation (DBS) in patients with early-stage Parkinson's disease (PD).

ELIGIBILITY:
Inclusion Criteria:

1. A clinical diagnosis of idiopathic Parkinson's disease (PD). The diagnosis will be based upon the presence of at least two of the three cardinal motor signs of this disorder (akinesia/bradykinesia, rest tremor, and rigidity) with at least one of the signs being rest tremor or bradykinesia.
2. Clear and dramatic beneficial response to dopaminergic therapy, defined as ≥30% in UPDRS III with administration of the patient's medication during the screening neurological examination.
3. Hoehn and Yahr (H&Y) stage II when OFF medication.
4. No contraindications to surgery (i.e., subject does not have uncontrollable medical or psychiatric illness; Exclusion Criteria).
5. Age between 50 and 75 years old.
6. Dopaminergic therapy for greater than one year and less than four years.
7. Available for follow-up for the entire duration of the study.
8. Informed Consent (Appendix C): The subject is willing and able to provide written informed consent.
9. MRI within normal range (Exclusion Criteria).
10. Subjects receiving antidepressant medication used specifically for the treatment of depression must be on stable doses for at least eight weeks prior to enrolling in the study.
11. Subjects must agree to maintain a stable regimen, if deemed medically appropriate by the treating physician, of any psychotropic medications throughout the blinded treatment phase.

Exclusion Criteria:

1. Evidence of an alternative diagnosis or secondary parkinsonism, as suggested by:

   * Features unusual early in the clinical course (e.g., prominent postural instability, freezing phenomena, or hallucinations unrelated to medications in the first 3 years after symptom onset)
   * Dementia preceding motor symptoms
   * Neurologic signs of upper motor neuron or cerebellar involvement
   * Significant orthostatic hypotension unrelated to medications
   * Unequivocal cortical sensory loss (i.e., graphesthesia, sterognosis with intact primary sensory modalities), clear limb ideomotor apraxia, or progressive aphasia
   * Vertical supranuclear gaze palsy, or selective slowing of vertical saccades
   * Unequivocal cerebellar abnormalities on examination, such as cerebellar gait, limb ataxia, or cerebellar oculomotor abnormalities (e.g., sustained gaze-evoked nystagmus, macro square wave jerks, hypermetric saccades)
   * Documentation of a condition known to produce parkinsonism and plausibly connected to the subject's symptoms (e.g., MRI scan with evidence of significant brain atrophy, lacunar infarcts, or iron deposits in the putamen; history of stroke, exposure to toxins, or encephalitis; or neuroleptic use within the past 6 months)
   * The expert evaluating physician, based on the full diagnostic assessment, believes that an alternative syndrome is more likely than PD.
2. Uncontrolled medical condition or clinically significant medical disease that would increase the risk of developing pre- or postoperative complications (e.g., significant cardiac or pulmonary disease, uncontrolled hypertension).
3. Dementia as evidenced by a Dementia Rating Score of less than 123.
4. Diagnosis of probable behavioral variant frontotemporal dementia or primary progressive aphasia.
5. Currently active diagnosis of a major psychiatric disorder.
6. Previous brain operation or injury.
7. Active participation in another clinical trial for the treatment of PD.
8. Subjects with cardiac pacemakers or medical conditions that require repeat MRI scans.
9. Evidence of existing dyskinesia
10. Any current substance use disorder.
11. Any history of recurrent or unprovoked seizures.
12. Any prior movement disorder treatments that involved intracranial surgery or device implantation.
13. Any other active implanted intracranial device (e.g., cochlear implant) or implanted device to treat movement disorders (e.g., duodopa pump) whether turned on or off.
14. A condition requiring or likely to require the use of magnetic resonance imaging (MRI) or diathermy.
15. History of suicide attempt.
16. A female who is breastfeeding or of child-bearing potential with a positive urine pregnancy test or not using adequate contraception.
17. Inability or unwillingness of subject to give written informed consent.
18. Parkinsonian features restricted to the lower limbs for more than three years.
19. Treatment with a dopamine receptor blocker or a dopamine-depleting agent in a dose and time course consistent with drug-induced parkinsonism.
20. Normal functional neuroimaging of the presynaptic dopaminergic system, as measured by DaTSCAN.
21. Rapid progression of gait impairment requiring regular use of a wheelchair.
22. Early bulbar dysfunction, defined as one of severe dysphonia, dysarthria (speech unintelligible most of the time), or dysphagia (requiring soft food, nasogastric (NG) tube, or gastrostomy feeding).
23. Inspiratory respiratory dysfunction defined as either diurnal or nocturnal inspiratory stridor or frequent inspiratory sighs.
24. Recurrent (>1/year) falls because of impaired balance within 3 years of onset.
25. Otherwise unexplained pyramidal tract signs, defined as pyramidal weakness or clear pathologic hyperreflexia (excluding mild reflex asymmetry in the more affected limb and isolated extensor plantar response).
26. Bilateral symmetric parkinsonism throughout the disease course. The patient or caregiver reports bilateral symptom onset with no side predominance, and no side predominance is observed on objective examination.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-08-30 (Estimated)

PRIMARY OUTCOMES:
frequency and severity of adverse events | 24 months
  frequency and severity of adverse events
frequency and severity of adverse cognitive outcome | 24 months
  decline from baseline at ≥ 1.5 SD (modest) and ≥ 2.0 (substantial) in tests comprising a comprehensive neuropsychological battery

SECONDARY OUTCOMES:
Stopped or Reversed Motor Progression | 24 months
  compare changes in motor progression for active DBS+ODT vs inactive DBS+ODT